CLINICAL TRIAL: NCT00170963
Title: Valsartan/Amlodipine 160/5 mg or 160/10 mg Versus Valsartan 160 mg Alone for 8 Weeks in Hypertensive Patients Who Are Not Adequately Controlled on Valsartan 160 mg Monotherapy
Brief Title: Efficacy and Safety of Valsartan/Amlodipine Combination in Hypertensive Patients Not Controlled With Valsartan Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAA489A2305
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Hypertension
Keywords: Hypertension, high blood pressure, valsartan, amlodipine
MeSH Terms: conditions — Hypertension | interventions — Amlodipine, Valsartan Drug Combination

INTERVENTIONS:
Drug: valsartan/amlodipine

SUMMARY:
This study will test the effectiveness and safety of a combination treatment in patients whose blood pressure is not controlled with a single medication

ELIGIBILITY:
Inclusion Criteria:

* Patients with uncomplicated, essential hypertension

Exclusion Criteria:

* Severe hypertension
* History of stroke, myocardial infarction, heart failure, chest pain, abnormal heart rhythm
* Liver, kidney, or pancreas disease
* Insulin dependent diabetes
* Allergy to certain medications used to treat high blood pressure

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 1018 (Actual)
Dates: Start 2004-10; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in diastolic blood pressure after 8 weeks

SECONDARY OUTCOMES:
Change from baseline in mean systolic blood pressure after 8 weeks
Decrease in diastolic blood pressure of at least 10 mmHg or diastolic blood pressure was less than 90 mmHg after 8 weeks
Diastolic blood pressure less than 90 mmHg after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Investigative Centers, Germany
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Derived] Sinkiewicz W, Glazer RD, Kavoliuniene A, Miglinas M, Prak H, Wernsing M, Yen J. Efficacy and tolerability of amlodipine/valsartan combination therapy in hypertensive patients not adequately controlled on valsartan monotherapy. Curr Med Res Opin. 2009 Feb;25(2):315-24. doi: 10.1185/03007990802630588. PMID 19192976